CLINICAL TRIAL: NCT07048002
Title: Interventions for Silent Brain Infarction and Perioperative Neurocognitive Disorders in Cardiovascular Surgery (the INSPIRE Study)
Brief Title: Interventions for Silent Brain Infarction and Perioperative Neurocognitive Disorders in Cardiovascular Surgery
Acronym: INSPIRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, SHI Jia, Vice Chair, Department of Anesthesiology, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: The INSPIRE study
Record Dates: First submitted 2025-06-12; First posted 2025-07-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-07

CONDITIONS: Silent Brain Infarction; Neurocognitive Disorders; Cardiac Surgery; Neuroprotective
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NeuroFirst target bundle (Experimental): Management for NeuroFirst target bundle
  Interventions: Other: Managements for NeuroFirst target bundle
- Routine Management (Active Comparator): Management for institutional routine in accordance with published guidelines
  Interventions: Other: Managements for institutional routine

INTERVENTIONS:
Other: Managements for NeuroFirst target bundle — In the intervention group, patient management aims to achieve the NeuroFirst target bundle, including 1) mean arterial pressure (MAP) 65-90 mmHg, 2) bispectral index (BIS) 40-60, 3) regional cerebral oxygen saturation (rSO2)≥ 60% , and 4) arterial inflow temperature <37 ℃ and rewarming rate < 0.5 ℃/min after exceeding 30℃ during CPB.
  To achieve this target bundle, pharmacologic agents, fluid resuscitation, blood transfusion, and other therapeutic modalities will be utilized. These interventions are guided by comprehensive intraoperative monitoring, including conventional hemodynamic monitoring, invasive or non-invasive cardiac output and vascular resistance assessments.
  Arms: NeuroFirst target bundle
Other: Managements for institutional routine — MAP, BIS, cerebral rSO2 and arterial inflow temperature during CPB rewarming, will be managed according to institutional routine in accordance with published guidelines.
  Arms: Routine Management

SUMMARY:
the purpose of the study is to investigate whether a combined anesthetic targets bundle, known as the NeuroFirst strategy, focused on neurological protection, can reduce the incidence of silent brain infarction (SBI) and perioperative neurocognitive disorders (PND) in patients undergoing cardiac surgery. Additionally, the trial will assess the safety of this strategy.

The NeuroFirst target bundle incorporates multiple parameters, including mean arterial pressure (MAP), bispectral index (BIS), regional cerebral oxygen saturation (rSO2), and arterial inflow temperature during cardiopulmonary bypass.

The primary question this study seeks to answer is: Does the NeuroFirst strategy reduce the incidence of SBI and PND in cardiac surgery?

To address this, researchers will compare the NeuroFirst strategy with routine institutional practices based on published guidelines. Participants will be randomly assigned to either the NeuroFirst group or the routine care group. All participants will undergo magnetic resonance imaging (MRI), be assessed using the Confusion Assessment Method (CAM) and the Montreal Cognitive Assessment (MoCA), and be followed for up to one year postoperatively.

ELIGIBILITY:
Inclusion criteria:

* Male or female adult patients aged 60 years or older
* Receiving elective cardiovascular surgery with cardiopulmonary bypass
* Written Informed consent provided

Exclusion criteria:

* Contraindication to MRI scanning
* Not suitable for receiving interventions to achieve NeuroFirst target bundle
* Unable to receive neuro-cognitive evaluation due to language, vision, or hearing impairments
* Breastfeeding or pregnancy
* Terminal illness with a life expectancy of less than 3 months
* Mental or legal disability
* current enrollment in other interventional study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 912 (Estimated)
Dates: Start 2025-07-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
the 7-day incidence of new-onset silent brain infarction (SBI) | within 7 days postoperatively
  New-onset silent brain infarction refers to newly developed cerebral infarctions detected on MRI, compared with the preoperative MRI, in the absence of any corresponding clinical symptoms of cerebral infarction.

SECONDARY OUTCOMES:
Key Secondary Outcome: the 30-day incidence of perioperative neurocognitive disorders (PND) | within 30 days postoperatively
  The incidence of 30-day PND includes the incidence of postoperative delirium in hospital and perioperative neurocognitive disorders within 30 days after surgery
the 5-day incidence of postoperative delirium | within five days postoperatively
  the incedence of delirium evaluated by CAM/CAM-ICU
the 30-day incidence of new-onset overt stroke | within 30 days postoperatively
  Postoperative new-onset overt stroke was defined as any new ischemic or hemorrhagic cerebrovascular event after surgery with focal or global neurological (motor, sensory or cognitive) dysfunction lasting at least 24 h. And a broadened stroke definition also including neurological dysfunction of <24 h duration with corresponding evidence of central nervous system hemorrhage or infarction (including pathological, imaging, or other objective evidence of cerebral, spinal cord or retinal focal ischemic injury in a defined vascular distribution).
the 1-year incidence of new-onset overt stroke | within 1 year postoperatively
  Postoperative new-onset overt stroke was defined as any new ischemic or hemorrhagic cerebrovascular event after surgery with focal or global neurological (motor, sensory or cognitive) dysfunction lasting at least 24 h. And a broadened stroke definition also including neurological dysfunction of <24 h duration with corresponding evidence of central nervous system hemorrhage or infarction (including pathological, imaging, or other objective evidence of cerebral, spinal cord or retinal focal ischemic injury in a defined vascular distribution).
the 1-year incidence of perioperative neurocognitive disorders (PND) | within 1 year postoperatively
  the incidence of perioperative neurocognitive disorders (PND)
the 30-day composite incidence of major adverse events | within 30 days postoperatively
  Major adverse events refer to renal insufficiency, myocardial infarction, pulmonary embolism, seizure and all-cause mortality.
the 1-year composite incidence of major adverse events | within 1 year postoperatively
  Major adverse events refer to renal insufficiency, myocardial infarction, pulmonary embolism, seizure and all-cause mortality.
the 30-day incidence of transient ischemic attack (TIA) | within 30 days postoperatively
  TIA is defined as focal arterial ischemia with transient symptoms (lasting <24 hours) and without evidence of infarction by pathology or imaging.
the 1-year incidence of transient ischemic attack (TIA) | within 1 year postoperatively
  TIA is defined as focal arterial ischemia with transient symptoms (lasting <24 hours) and without evidence of infarction by pathology or imaging.

OTHER OUTCOMES:
Length of stay (LOS) in intensive care unit (ICU) | Perioperative
  Length of stay (LOS) in intensive care unit (ICU) postoperatively
Length of stay (LOS) in hospital | Perioperative
  Length of stay (LOS) in hospital postoperatively
Hospitalization cost | Perioperative
  Operative and postoperative hospitalization cost

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Beijing Chaoyang Hospital，Capital Medical University, Beijing, Beijing Municipality
  - State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences & Peking Union Medical College, Beijing, Beijing Municipality
  - Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The Central Hospital of Wuhan, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared in order to protect participant privacy and confidentiality. Additionally, the consent obtained from participants does not include provisions for data sharing, in accordance with ethical guidelines and institutional policies.

REFERENCES:
- [Background] Uysal S, Lin HM, Trinh M, Park CH, Reich DL. Optimizing cerebral oxygenation in cardiac surgery: A randomized controlled trial examining neurocognitive and perioperative outcomes. J Thorac Cardiovasc Surg. 2020 Mar;159(3):943-953.e3. doi: 10.1016/j.jtcvs.2019.03.036. Epub 2019 Mar 29. PMID 31056357
- [Background] Maheshwari A, McCormick PJ, Sessler DI, Reich DL, You J, Mascha EJ, Castillo JG, Levin MA, Duncan AE. Prolonged concurrent hypotension and low bispectral index ('double low') are associated with mortality, serious complications, and prolonged hospitalization after cardiac surgery. Br J Anaesth. 2017 Jul 1;119(1):40-49. doi: 10.1093/bja/aex095. PMID 28974062
- [Background] Descamps R, Amour J, Besnier E, Bougle A, Charbonneau H, Charvin M, Cholley B, Desebbe O, Fellahi JL, Frasca D, Labaste F, Lena D, Mahjoub Y, Mertes PM, Molliex S, Moury PH, Moussa MD, Oilleau JF, Ouattara A, Provenchere S, Rozec B, Parienti JJ, Fischer MO; OPTIPAM investigators. Perioperative individualized hemodynamic optimization according to baseline mean arterial pressure in cardiac surgery patients: Rationale and design of the OPTIPAM randomized trial. Am Heart J. 2023 Jul;261:10-20. doi: 10.1016/j.ahj.2023.03.005. Epub 2023 Mar 18. PMID 36934980
- [Background] Gerstenecker A, Norling AM, Jacob A, Lazar RM. Silent Brain Infarction, Delirium, and Cognition in Three Invasive Cardiovascular Procedures: a Systematic Review. Neuropsychol Rev. 2023 Jun;33(2):474-491. doi: 10.1007/s11065-022-09548-1. Epub 2022 Jul 8. PMID 35804216
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Brown CH 4th, Probert J, Healy R, Parish M, Nomura Y, Yamaguchi A, Tian J, Zehr K, Mandal K, Kamath V, Neufeld KJ, Hogue CW. Cognitive Decline after Delirium in Patients Undergoing Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):406-416. doi: 10.1097/ALN.0000000000002253. PMID 29771710
- [Background] Cheng C, Wan H, Cong P, Huang X, Wu T, He M, Zhang Q, Xiong L, Tian L. Targeting neuroinflammation as a preventive and therapeutic approach for perioperative neurocognitive disorders. J Neuroinflammation. 2022 Dec 12;19(1):297. doi: 10.1186/s12974-022-02656-y. PMID 36503642
- [Background] Indja B, Woldendorp K, Vallely MP, Grieve SM. Silent Brain Infarcts Following Cardiac Procedures: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2019 May 7;8(9):e010920. doi: 10.1161/JAHA.118.010920. PMID 31017035
- [Background] Vermeer SE, Prins ND, den Heijer T, Hofman A, Koudstaal PJ, Breteler MM. Silent brain infarcts and the risk of dementia and cognitive decline. N Engl J Med. 2003 Mar 27;348(13):1215-22. doi: 10.1056/NEJMoa022066. PMID 12660385
- [Background] Fanning JP, Wong AA, Fraser JF. The epidemiology of silent brain infarction: a systematic review of population-based cohorts. BMC Med. 2014 Jul 9;12:119. doi: 10.1186/s12916-014-0119-0. PMID 25012298
- [Background] Sultan I, Bianco V, Kilic A, Jovin T, Jadhav A, Jankowitz B, Aranda-Michel E, D'angelo MP, Navid F, Wang Y, Thoma F, Gleason TG. Predictors and Outcomes of Ischemic Stroke After Cardiac Surgery. Ann Thorac Surg. 2020 Aug;110(2):448-456. doi: 10.1016/j.athoracsur.2020.02.025. Epub 2020 Mar 19. PMID 32199830